CLINICAL TRIAL: NCT07382596
Title: Cervical Plexus Hydrodissection With D5W Versus NS for Treatment-Resistant PTSD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Dean Reeves Clinic (Other)
Responsible Party: Principal Investigator, Dr. Dean Reeves, Principal Investigator, Dr. Dean Reeves Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCPHD-D5WvsNSforPTSD
Record Dates: First submitted 2026-01-24; First posted 2026-02-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: PTSD
Keywords: Dextrose; Hydrodissection; Cervical Plexus
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: Randomized double-blind study comparing BHDCP with D5W versus NS
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The statistician is masked as well
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- D5W cervical plexus hydrodissection (Experimental): 10 ml D5W cervical plexus hydrodissection bilaterally at 0, 2, 4, and 8 weeks, and then by request from 13-52 weeks
  Interventions: Drug: Dextrose 5% in water bilateral injection
- Normal saline cervical plexus hydrodissection (Active Comparator): 10 mL normal saline cervical plexus hydrodissection bilaterally at 0, 2, 4, and 8 weeks, and then D5W by request from 13-52 weeks
  Interventions: Drug: Normal saline bilateral injection

INTERVENTIONS:
Drug: Dextrose 5% in water bilateral injection — Injection under the investing fascia of the sternocleidomastoid muscle
  Arms: D5W cervical plexus hydrodissection
Drug: Normal saline bilateral injection — Injection under the investing fascia of the sternocleidomastoid muscle
  Arms: Normal saline cervical plexus hydrodissection

SUMMARY:
PTSD is a chronic mental health condition that drastically reduces an individual's quality of life Dextrose injection with a small needle has been used for chronic pain patients and observational results have shown it to be effective in reducing anxiety, brain fog, and depression in patients with PTSD. This randomized trial will compare dextrose injection with an injection control of normal saline (NS)

DETAILED DESCRIPTION:
PTSD is a well-recognized debilitating mental health condition associated with previous trauma exposure. It is part of the DSM-5 Trauma and Stressor related disorders category. Treatments for PTSD normally involve a multi-disciplinary approach. First-line treatments include psychotherapy and serotonergic reuptake inhibitors. Many patients fail pharmacotherapy and psychotherapy. Unilateral stellate ganglion block performed favorably for treatment of PTSD in a recent RCT, based upon an expectation that the cervical sympathetic system is neuropathically upregulated in PTSD. However, inclusion of lidocaine requires the presence of an emergency response team due to the potential for inadvertent intravascular injection with generalized seizures or hypotension, and inadvertent laryngeal or phrenic nerve block. Perineural injection of peripheral nerves, plexi, or sympathetic ganglia with dextrose 5% in water (D5W), has performed well empirically in the treatment of post-traumatic stress disorder. No lidocaine is utilized, which allows for avoidance of lidocaine toxicity risk, or any risk of nerve block. Because of that, bilateral procedures are feasible, and these procedures can be performed in any outpatient office with ultrasound availability, as emergency team backup is not necessary, making the procedure readily accessible. A cumulative benefit has been observed, as well. The effects of BHDCP with D5W as a stand-alone treatment for PTSD is under evaluated in a randomized trial compared treatment with D5W versus delayed treatment with early results promising. This study is designed as the next step in study quality through use of an injection control. The primary outcome is the short term and long-term effect of BHDCP with D5W versus NS on the Post Traumatic Stress Disorder Check List for Civilians (PCL-C), The primary hypotheses are tha cervical plexus hydrodissection with D5W will outperform NS for the primary measure, and that the PCL_C improvement will be equal to or greater than 15.3 (1.5 times the MCID of 10.2.). A study size of 50 planned, based on power analysis.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* Not involved in another study of PTSD treatment
* Reliable transportation
* Comfortable with computers
* Tried 2 or more medications for treatment of PTSD symptoms
* Tried 2 or more non-medication treatments for PTSD symptom
* No known life-threatening illness
* Not taking daily narcotics
* Not having 3 or more alcoholic drinks on an average day
* No active suicidal plans
* No major surgery plans
* No major life stress that might interfere with completing study
* Symptoms for more than 1 year
* Not planning to move for next 18 months.
* Living within an hour of Portland, OR, Madison, WI, or Lexington, KY
* Wiling to provide 2 email and 2 phone contact methods
* Willing to answer questions on multiple occasions over the course of a year.
* Willing to be assigned to 3 months of usual care treatment
* No diagnosis of schizophrenia, Borderline Personality Disorder, or Bipolar Disorder.
* No severe needle phobia
* Chronic pain ≤ 5/10
* PCL-C score ≥ 50

Exclusion Criteria:

-

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Post traumatic checklist for civilians | 3 months
  Minimum 17 Maximum 85 Higher scores mean worse outcome

SECONDARY OUTCOMES:
Hospital anxiety and depression scale | 3 months
  Minimum 0 Maximum 42 Higher scores mean worse outcome
EuroQol Visual Analog Scale (0-100 overall quality of life) | 3 months
  Minimum 0 Maximum 100 Higher scores mean better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth D Reeves, M.D., Principal Investigator — Dr. Dean Reeves Clinic
Locations (4):
- United States (4):
  - Wellward Medical, Lexington, Kentucky
  - NW Regen, Portland, Oregon
  - Paul Johnson, MD., Portland, Oregon
  - Medical Procedures of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
De-identified data are available from the first author upon request in writing and with a detailed use plan.
Time Frame: 10 years
Access Criteria: Request in writing